CLINICAL TRIAL: NCT06229483
Title: The Effects of Intraoperative Tranexamic Acid on Perioperative Bleeding In Craniotomies
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stephen Lownie (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Stephen Lownie, Professor, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TXA-2024-01
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Brain Tumor; Bleeding
MeSH Terms: conditions — Brain Neoplasms; Hemorrhage | interventions — Tranexamic Acid; Injections, Intravenous; Solutions; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive a 20 mg/kg IV bolus of TXA, or identical volume of placebo 0.9 % NaCl will be administered intravenously push by the anesthesiologist approximately 30 minutes prior to the skin incision followed by a 1 mg/kg/hr infusion of TXA, or identical volume of placebo 0.9 % NaCl, for the duration of surgery
Who Masked: Participant
Masking Description: This is a blinded study. The participant, surgeon and research team will not know the treatment allocation. Only the pharmacy preparing the medication will be unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Experimental): Participants will be randomized in a 1:1 ratio to receive tranexamic acid 20 mg/kg IV bolus or identical volume of placebo 0.9 % NaCl within 30 minutes prior to the skin incision followed by a 1 mg/kg/hr infusion of TXA, or identical volume of placebo 0.9 % NaCl, for the duration of surgery. Treatment is blinded.
  Interventions: Drug: TRANEXAMIC ACID 1 G in 10 mL INTRAVENOUS INJECTION, SOLUTION
- Matching Placebo (Placebo Comparator): Participants will be randomized in a 1:1 ratio to receive tranexamic acid 20 mg/kg IV bolus or identical volume of placebo 0.9 % NaCl within 30 minutes prior to the skin incision followed by a 1 mg/kg/hr infusion of TXA, or identical volume of placebo 0.9 % NaCl, for the duration of surgery. Treatment is blinded.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TRANEXAMIC ACID 1 G in 10 mL INTRAVENOUS INJECTION, SOLUTION — Tranexamic acid 20 mg/kg IV bolus within 30 minutes prior to the skin incision followed by a 1 mg/kg/hr infusion of TXA, for the duration of surgery. Treatment is blinded.
  Other Names: TXA
  Arms: Tranexamic Acid
Other: Placebo — 0.9% normal saline 20ml/kg IV bolus within 30 minutes prior to the skin incision followed by a 1 ml/kg/hr infusion of 0.9 % sodium chloride for the duration of surgery. Treatment is blinded.
  Other Names: Normal saline (0.9% sodium chloride)
  Arms: Matching Placebo

SUMMARY:
The goal of this clinical trial is to test the effect of a drug called tranexamic acid (TXA) on reducing blood loss in participants undergoing surgery to remove brain tumors. The main questions it aims to answer are:

1. Does TXA 20 mg/kg IV bolus of TXA, and 1 mg/kg/hr infusion of TXA reduce the amount of estimated blood loss during surgery?
2. Does TXA 20 mg/kg IV bolus of TXA, and 1 mg/kg/hr infusion of TXA prevent re-operation, disability or death related to bleeding inside the head during and after surgery? Participants are randomized to receive 20 mg/kg IV bolus of TXA or matching placebo within 30 minutes of start of surger, and then 1 mg/kg/hr infusion of TXA or matching from the start of surgery to end of surgery. Treatment allocation is blinded. Investigator will compare the two treatment arms to see whether there are differences in the amount of blood loss during surgery and bleeding-related complications. Investigators will also monitor for any side effects of TXA.

DETAILED DESCRIPTION:
Excessive blood loss during and after a neurosurgical procedure may increase illness and cause death. The surgeons and their team put in a lot of effort during surgery to and prevent excessive bleeding during and after surgery. One of the medications that may help is tranexamic acid (TXA). TXA is a medication that is widely used in cardiac, orthopedic and trauma surgery to prevent heavy bleeding, the need for blood transfusion and reduce death. During neurosurgery, there is not enough proof whether giving TXA to participants reduces blood loss, and there are no clear guidelines regarding the use of TXA. Investigators are interested in studying the effect of TXA on blood loss in participants undergoing craniotomy to remove a brain tumor. A craniotomy is an operation where a piece of the skull is removed to show part of the brain to remove a brain tumor. One of the risks associated with this procedure is bleeding. Currently, some participants undergoing this type of surgery receive TXA and others do not, as the decision to administer TXA is based on an investigator's preference. Therefore, a study investigating the impact of TXA on bleeding during or following craniotomy, as well as its safety, is needed to better inform practice and potentially improve outcomes of surgery.

ELIGIBILITY:
Inclusion Criteria are the following:

1. Adult male or female, between 18-80 years of age.
2. Patients are scheduled to undergo a craniotomy for tumor resection.
3. Patients/ Substitute Decision Maker have given written consent to participate.

Exclusion Criteria are the following: Patients who meet any of the following exclusion criteria will not be eligible.

1. Patients with known active or previous history of thromboembolic disease or deep venous thrombosis.
2. Patients with known pre-existing coagulopathy such as hemophilia, Von Willebrand disease, and clotting factor deficiencies.
3. Patients with renal impairment and eGFR <60 ml/min/1.73 m2 as determined by the lab or calculated by using the Cockcroft Gault formula or end stage renal disease currently on dialysis.
4. Female subjects who are pregnant or currently breastfeeding.
5. Patients with Class 3 (high-risk) obesity BMI ≥ to 40.
6. Patients undergoing emergency craniotomy or mini craniotomy or craniectomies.
7. Patients who received embolization prior to surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimated intraoperative blood loss | Surgery
  a. EBL (ml/kg) = ERCV lost (ml)/[weight (kg) x hematocrit preop/100] i. ERCV = EBV x hematocrit/100 ii. ERCV lost = ERCV preop + ERCV transfused - ERCV postop iii. ERCV transfused = PRBC transfused (ml) x hematocrit transfused PRBC/100 iv. EBV = 75 ml/kg x weight (kg) b. abbreviations used: EBL, estimated blood loss; ERCV, estimated red cell volume; EBV, estimated blood volume; PRBC, packed red blood cells
Reoperation or disability or death due to intracranial hemorrhage within 30 days | 30 days

SECONDARY OUTCOMES:
What is the difference in Hemoglobin level postoperatively as compared to baseline? | 24 hrs
Number of subjects requiring transfusion of blood products | 30 days
Volume of transfused packed red blood cell (PRBC) and fresh frozen plasma (FFP) | 30 days
What is the difference in Intraoperative hemodynamics between subjects? | Surgery
Length of operation | Surgery
Length of intensive care unit (ICU)/hospital stay | 30 days
Medication related risks, including seizure, thromboembolic event | 30 days
What is the difference in Platelet level postoperatively as compared to baseline? | 24 hrs
What is the difference in Fibrinogen level postoperatively as compared to baseline? | 24 hrs
What is the difference in INR/PTT value level postoperatively as compared to baseline? | 24 hrs
What is the difference in Hematocrit level postoperatively as compared to baseline? | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lownie, MD, Principal Investigator — Nova Scotia Health Authority- Queen Elizabeth II HSC
Locations (1):
- Nova Scotia Health Authority- Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rajagopalan V, Chouhan RS, Pandia MP, Lamsal R, Rath GP. Effect of Intraoperative Blood Loss on Perioperative Complications and Neurological Outcome in Adult Patients Undergoing Elective Brain Tumor Surgery. J Neurosci Rural Pract. 2019 Oct;10(4):631-640. doi: 10.1055/s-0039-3399487. Epub 2019 Dec 11. PMID 31831982
- [Result] Rolston JD, Han SJ, Lau CY, Berger MS, Parsa AT. Frequency and predictors of complications in neurological surgery: national trends from 2006 to 2011. J Neurosurg. 2014 Mar;120(3):736-45. doi: 10.3171/2013.10.JNS122419. Epub 2013 Nov 22. PMID 24266542
- [Result] Hooda B, Chouhan RS, Rath GP, Bithal PK, Suri A, Lamsal R. Effect of tranexamic acid on intraoperative blood loss and transfusion requirements in patients undergoing excision of intracranial meningioma. J Clin Neurosci. 2017 Jul;41:132-138. doi: 10.1016/j.jocn.2017.02.053. Epub 2017 Mar 7. PMID 28283245
- [Result] Vel R, Udupi BP, Satya Prakash MV, Adinarayanan S, Mishra S, Babu L. Effect of low dose tranexamic acid on intra-operative blood loss in neurosurgical patients. Saudi J Anaesth. 2015 Jan;9(1):42-8. doi: 10.4103/1658-354X.146304. PMID 25558198
- [Result] Eustache G, Nardi N, Rousseau C, Aouaissia S, Aillet S, Delahaye Larralde S, Wodey E, Riffaud L. Importance of tranexamic acid in pediatric monosutural craniosynostosis surgery. J Neurosurg Pediatr. 2021 Dec 24;29(4):412-418. doi: 10.3171/2021.10.PEDS21438. Print 2022 Apr 1. PMID 34952528
- [Result] Crantford JC, Wood BC, Claiborne JR, Ririe DG, Couture DE, Thompson JT, David LR. Evaluating the safety and efficacy of tranexamic acid administration in pediatric cranial vault reconstruction. J Craniofac Surg. 2015 Jan;26(1):104-7. doi: 10.1097/SCS.0000000000001271. PMID 25534062
- [Result] Wu B, Lu Y, Yu Y, Yue H, Wang J, Chong Y, Cui W. Effect of tranexamic acid on the prognosis of patients with traumatic brain injury undergoing craniotomy: study protocol for a randomised controlled trial. BMJ Open. 2021 Nov 25;11(11):e049839. doi: 10.1136/bmjopen-2021-049839. PMID 34824110
- [Result] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Result] Brown NJ, Hartke JN, Pacult M, Burkett KR, Gendreau J, Catapano JS, Lawton MT. Tranexamic Acid Demonstrates Efficacy without Increased Risk for Venous Thromboembolic Events in Cranial Neurosurgery: Systematic Review of the Evidence and Current Applications in Nontraumatic Pathologies. World Neurosurg. 2024 Mar;183:29-40. doi: 10.1016/j.wneu.2023.11.148. Epub 2023 Dec 3. PMID 38052364